CLINICAL TRIAL: NCT02800421
Title: Prognostic Impact of Combined Contrast-Induced Acute Kidney Injury and Hypoxic Liver Injury in Patients With ST Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Prognostic Impact of Organ Damage in STEMI Patients
Status: Completed | Type: Observational
Sponsor: Inha University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INHAUH 2016-05-015
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Myocardial Infarction; Death; Acute Kidney Injury; Hepatic Insufficiency
MeSH Terms: conditions — Myocardial Infarction; Death; Acute Kidney Injury; Hepatic Insufficiency

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- no organ damage: no evidence of HLI and CI-AKI
- CI-AKI only: CI-AKI, but no HLI
- HLI only: HLI, but no CI-AKI
- combined CI-AKI and HLI: Both CI-AKI and HLI

SUMMARY:
Besides contrast-induced acute kidney injury (CI-AKI), adscititious vital organ damage such as hypoxic liver injury (HLI) may affect the survival in patients with ST-elevation myocardial infarction (STEMI). Therefore, the investigator sought to evaluate the prognostic impact of CI-AKI and HLI in STEMI patients who underwent primary percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
A total of 668 consecutive patients (77.2% male, mean age 61.3±13.3 years) with STEMI underwent primary PCI were analyzed. Hypertension was defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg, or by antihypertensive prescription. Type 2 diabetes was defined by hypoglycemic agents or insulin prescription, fasting plasma glucose ≥126 mg/dL, glycosylated hemoglobin (HbA1c) ≥6.5%, or known but untreated hyperglycemia. Dyslipidemia was defined by total cholesterol ≥240 mg/dL, LDL cholesterol ≥130 mg/dL, HDL cholesterol<40 mg/dL, triglycerides ≥200 mg/dL, and/or by lipid-lowering prescription.STEMI was defined as typical chest pain lasting for >30 min within the last 24h, with electrocardiographic findings of ST elevation >1 mm in at least two consecutive leads or new-onset left bundle branch block, and 2-fold elevation of serum levels of troponin-I or the creatine kinase-MB above the upper normal limit. Obstructive CAD was defined as ≥50% luminal narrowing and the extent of obstructive CAD was categorized according to the number of vessels involved (1, 2, or 3). CI-AKI was defined as increase in serum creatinine of ≥0.5 mg/dl or 25% relative rise, within 48h after index procedure. HLI was defined as ≥2-fold increase of serum aspartate transaminase above upper normal limit at admission. Patients were divided into four groups according to their CI-AKI and HLI states. Major adverse cardiovascular and cerebrovascular events (MACCE) defined as composite of all-cause mortality, non-fatal MI, non-fatal stroke, ischemia-driven target lesion revascularization and target vessel revascularization were recorded. Continuous data were expressed as a mean value ± standard deviation or median value (interquartile range) as appropriate. Categorical data were presented as a percentage or absolute number. Analyses of continuous data were performed using analysis of variance (ANOVA) test or Kruskal-Wallis test as appropriate and analyses of categorical data were performed using chi-square test to assess differences among the four groups. Cumulative event rates as a function over time were estimated using the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients who undergone primary PCI

Exclusion Criteria:

* Chronic liver disease
* Life expectancy < 1year

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 668 STEMI patients (77.2% male, mean age 61.3±13.3 years) with STEMI underwent primary PCI between 2007 and 2014 were enrolled. Primary PCI was performed according to standard clinical practice. Pharmacological therapy, temporary pacemaker insertion, and intra-aortic balloon pump support were left to the operators' discretion.
Sampling Method: Non-Probability Sample
Enrollment: 668 (Actual)
Dates: Start 2007-01; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
composite major adverse cardiovascular and cerebrovascular event (MACCE) | an average of 2 years
  all-cause mortality, non-fatal MI, non-fatal stroke, and ischemia-driven TLR/TVR

IPD SHARING:
Plan to Share IPD: Undecided
Sharing individual participant data is available, since I have full data encoded. However, if it is feasible uploading the individual data, I would consider it positively.

REFERENCES:
- [Derived] Choi SH, Jang HJ, Suh YJ, Park SD, Oh PC, Moon J, Lee K, Suh J, Kang W, Kim TH, Kwon SW. Clinical Implication of Hypoxic Liver Injury for Predicting Hypoxic Hepatitis and In-Hospital Mortality in ST Elevation Myocardial Infarction Patients. Yonsei Med J. 2021 Oct;62(10):877-884. doi: 10.3349/ymj.2021.62.10.877. PMID 34558866
- [Derived] Park SD, Moon J, Kwon SW, Suh YJ, Kim TH, Jang HJ, Suh J, Park HW, Oh PC, Shin SH, Woo SI, Kim DH, Kwan J, Kang W. Prognostic Impact of Combined Contrast-Induced Acute Kidney Injury and Hypoxic Liver Injury in Patients with ST Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention: Results from INTERSTELLAR Registry. PLoS One. 2016 Jul 14;11(7):e0159416. doi: 10.1371/journal.pone.0159416. eCollection 2016. PMID 27415006